CLINICAL TRIAL: NCT06092333
Title: A Pilot Study of the Combination of VIR-2218 and Peginterferon Alfa-2a for Chronic Hepatitis B
Brief Title: VIR-2218 and Peginterferon Alfa-2a for Chronic Hepatitis B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001606; 001606-DK
Record Dates: First submitted 2023-10-19; First posted 2023-10-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-13

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Treatment; Functional Cure; Immune Response
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm, open label (Other): open label
  Interventions: Drug: VIR-2218 and peginterferon alfa-2a

INTERVENTIONS:
Drug: VIR-2218 and peginterferon alfa-2a — (VIR-2218) administered as a lead-in followed by combination with peginterferon alfa-2a

SUMMARY:
Background:

Chronic hepatitis B virus (HBV) infection affects 292 million people worldwide; 887,000 die each year from cirrhosis, liver cancer, and related issues. Treatment options are limited.

Objective:

To test 2 drugs (VIR-2218 and peginterferon) in people with mild or inactive HBV infection.

Eligibility:

People aged 18 to 65 years with mild or inactive HBV infection.

Design:

Participants will be screened. They will have blood tests and an eye exam. They will have imaging scans of the liver to check the health of the liver.

Participants will be in the study for over 2 years.

VIR-2218 is an injection given under the skin of the stomach, upper arm, or thigh. Participants will come to the clinic to receive this injection once a month for 6 months.

Peginterferon is also injected under the skin. Participants will have this shot once a week for 6 months. They may either inject themselves at home or come to the clinic to get the injections.

Participants will get just the VIR-2218 for 3 months, then both shots for 3 months, then just the peginterferon for 3 months.

Participants will have two 3-day stays in the hospital. Tests will include:

Liver biopsy. A sample of tissue will be taken from their liver. After the procedure, participants will lie on their right side for 2 hours and then on their back for 4 hours.

Fine needle aspiration. A small needle will be used to collect cells from the liver.

After the last injection of peginterferon, follow-up visits will continue in the outpatient clinic every 4 to 12 weeks.

DETAILED DESCRIPTION:
Study Description:

Up to 50 untreated, adult, male and female subjects with hepatitis B e antigen (HBeAg) negative chronic hepatitis B (CHB) with low level viremia and antigenemia (hepatitis B surface antigen (HBsAg)) without cirrhosis will be screened in order to enroll 10 subjects in an open-label, phase 2a, single site (NIH Clinical Center), single arm, proof-of-concept study of a siRNA (VIR-2218) administered as a lead-in followed by combination with peginterferon alfa-2a. The primary endpoint of the study is log decline in quantitative HBsAg (qHBsAg) level. Secondary objectives include safety, functional cure defined as undetectable HBsAg (<low limit of detection (LLOD) 0.085 IU/ml) and sustained suppression of HBV DNA [<lower limit of quantification (LLOQ]) <10 IU/ml)] 24 weeks after discontinuation of all treatment (study week 60), antiviral activity, and to understand immunological changes following reduction/removal of HBsAg and to evaluate novel markers to monitor treatment response. A tertiary objective will be to assess the durability of the primary endpoint at week 120 (84 weeks after stopping treatment). After screening, eligible subjects will undergo a baseline liver biopsy followed by subcutaneous (SC) administration of VIR-2218 every 4 weeks followed by a repeat liver biopsy at week 12. Thereafter, peginterferon alfa-2a 180 ug mcg SC weekly will be initiated in combination with VIR-2218 for 12 weeks followed by peginterferon alfa-2a alone weekly for another 12 weeks. Total treatment duration will be 36 weeks (6 doses of VIR-2218 and 24 doses of peginterferon alfa-2a). Fine needle aspirates of the liver and blood for peripheral blood mononuclear cells (PBMCs) will be collected throughout the study to assess intrahepatic and peripheral immune parameters, respectively.

Objectives:

Primary Objective

1. To evaluate the effect of administration of VIR-2218 in combination with peginterferon alfa-2a on qHBsAg levels

Secondary Objectives

1. To evaluate the safety and tolerability of VIR-2218 in combination with peginterferon alfa-2a in non-cirrhotic adults with chronic HBV infection
2. To evaluate functional cure following administration of VIR-2218 in combination with peginterferon alfa-2a
3. To evaluate the antiviral activity of VIR-2218 in combination with peginterferon alfa-2a in non-cirrhotic adults with chronic hepatitis B virus (HBV) infection.
4. To evaluate the effects of VIR-2218 in combination with peginterferon alfa-2a on peripheral and intrahepatic immune responses in non-cirrhotic adults with chronic HBV infection
5. To evaluate for the development of antiviral resistance during administration of VIR-2218 in combination with peginterferon alfa-2a

Exploratory Objectives

1. To evaluate other markers of HBV infection
2. To evaluate potential biomarkers for host responses to infection and/or to therapy
3. To compare intrahepatic and peripheral immune response obtained by fine needle aspiration (FNA) and PBMC, respectively
4. To assess the durability of the primary endpoint at week 120 (84 weeks after all treatment is discontinued)

Endpoints:

Primary Endpoint

1. Decline in log IU/mL quantitative HBsAg level 24 weeks after discontinuation of all treatment (study week 60)

Secondary Endpoints

1. Safety
2. Functional cure which is defined as undetectable HBsAg (<0.085 IU/ml) AND sustained suppression of HBV DNA [< LLOQ], <10 IU/ml)] for more than 6 months after discontinuation of all treatment
3. HBV DNA <10 IU/ml at end of treatment and 6 months off treatment. The response will be reported as HBV DNA <LLOQ target detected (TD) or target not detected (TND)
4. Changes in innate and adaptive host immune responses to HBV during and after treatment.

   * Greater natural killer (NK) cell response to the first peginterferon injection (measured as increase in TNFrelated apoptosis-inducing ligand (TRAIL)-expressing natural killer (NK) cell within the first 6 hours after peginterferon injection) in patients in this study compared to historic control
   * Preferential improvement of HBsAg-specific T cell responses (measured as increase in the frequency of interferon gamma (IFN-g) producing T cells from baseline to week 12, from baseline to week 36 and from baseline to week 84) as compared to HBV core and polymerasespecific T cell responses in the same patients.

Tertiary Endpoints

1. HBV RNA, hepatitis B core-related antigen (HBcrAg), HBV DNA by digital droplet polymerase chain reaction (ddPCR)
2. qHBsAg using an ultrasensitive assay with a LLOQ of 0.005 IU/mL
3. Analysis of stool samples for microbiota (16s rRNA gene sequencing), Fibroscan.
4. Exploratory analysis of additional immunological parameters in serum, blood and liver and/or use of additional analysis techniques to further our understanding of changes in immune function during/after treatment.
5. To assess the durability of the primary endpoint at week 120 (84 weeks after all treatment is discontinued)

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age >=18-65 years
2. HBsAg positive with a level <2,000 IU/mL at the time of screening
3. Hepatitis B e antigen negative
4. HBV DNA levels <10,000 IU/mL on two occasions at least 24 weeks apart with the second being at time of screening
5. ALT level <=2 ULN (using sex-specific cut-offs of normal 35 U/L for males and 25 U/L for females) based on at least two determinations taken at least 24 weeks apart with the second being at time of screening

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or lactation
2. For women of childbearing potential, inability, or unwillingness to use highly effective contraception during study drug dosing and for an additional 24 weeks after the end of study drug administration.
3. For males of reproductive potential: Unable or unwilling to use condoms consistently in addition to female partner using another adequate contraceptive method to ensure effective contraception with partner during study participation and for an additional 24 weeks after the end of study medication administration. Patients who have underwent surgical sterilization (vasectomy) will still require female partner to utilize an additional adequate contraception method.
4. Known history of hypersensitivity or contraindication to an siRNA, oligonucleotide, or GalNAc or any interferon product
5. Current use of oral theophylline and methadone
6. Any treatment for HBV within the last 24 weeks
7. Prior exposure to a siRNA
8. Co-infection with HDV as defined by the presence of anti-HDV in serum.
9. Co-infection with HCV as defined by the presence of anti-HCV and HCV RNA in serum.
10. Co-infection with HIV as defined by the presence of anti-HIV in serum
11. Cirrhosis either diagnosed by a prior liver biopsy at any time or, if not available, by a transient elastography score >13 kPa
12. Decompensated liver disease as defined by serum bilirubin >2.5 mg/dL (with direct bilirubin > 1.5 mg/dL), prothrombin time of greater than 2 seconds prolonged, a serum albumin of less than 3.5 g/dL, or a history of ascites, variceal bleeding or hepatic encephalopathy
13. Hepatocellular carcinoma (HCC), or the presence of a mass on imaging studies of the liver that is suggestive of HCC, or an alpha-fetoprotein level of greater than 500 ng/mL
14. Presence of other causes of liver disease, (i.e. hemochromatosis, Wilson disease, alcoholic liver disease, severe steatosis, alpha-1-anti-trypsin deficiency)
15. A history of solid organ or bone marrow transplant
16. Any current medical condition requiring the chronic use of more than 10 mg of prednisone (or its equivalent) daily or biologics (e.g. monoclonal antibody, interferon) within 3 months of screening.
17. Significant systemic illness other than liver diseases including congestive heart failure, renal failure, chronic pancreatitis and diabetes mellitus with poor control (hemoglobin A 1C (HgbA1C >8.5)), that in the opinion of the investigator may interfere with therapy.
18. eGFR < 60 ml/min, serum creatinine > 1.3 mg/dl
19. Platelet count <90 mm3/dL
20. Hgb <12 g/dL for males and <11 g/dL for females
21. White Blood cell count < 2500 cells/mm3
22. Neutrophil count < 1500 cell/mm3 (or < 1000 cell/mm3 if considered a physiological variant in a subject of African descent)
23. Active ethanol/drug abuse/psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, or personality disorder that, in the investigator s opinion, might interfere with participation in the study.
24. History of malignancy or treatment for a malignancy within the past 3 years (except adequately treated carcinoma in situ or basal cell carcinoma of the skin).
25. History of immune-mediated disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune hepatitis, sarcoidosis, psoriasis of greater than mild severity, autoimmune uveitis), or cerebrovascular, chronic pulmonary or cardiac disease associated with functional limitation, retinopathy, uncontrolled thyroid disease, (TSH >10 or <0.4mU/L) or uncontrolled seizure disorder, as determined by a study physician.
26. Use of another investigational agent within 90 days of screening
27. Use of any prohibited immunosuppressants (except short term use of prednisone as a steroid burst [<= 1 week of use]) or cytotoxic medications
28. Presence of conditions that, in the opinion of the investigators, would not allow the patient to be followed in the current study.
29. Inability of subject to understand and the unwillingness to sign a written informed consent document

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Decline in log quantitative HBsAg level | 6 months after discontinuation of all treatment
  To evaluate the effect of administration of VIR-2218 in combination with peginterferon alfa-2a on qHBsAg levels

SECONDARY OUTCOMES:
Changes in innate and adaptive host immune responses to HBV during and after treatment. | Within the first 6 hours after peginterferon injection; Baseline to week 12, from Baseline to week 36 and from Baseline to week 84
  To evaluate the effects of VIR-2218 in combination with peginterferon alfa-2a on peripheral and intrahepatic immune responses in non-cirrhotic adults with chronic HBV infection
HBV DNA <10 IU/ml at end of treatment and 6 months off treatment. The response will be reported as HBV DNA <LLOQ target detected (TD) or target not detected (TND) | 6 months off-treatment
  Partial cure. An alternative goal of treatment of chronic hepatitis B
Functional cure which is defined as undetectable HBsAg (<0.085 IU/ml) AND sustained suppression of HBV DNA [< LLOQ], <10 IU/ml)] for more than 6 months after discontinuation of all treatment | > 6 months after discontinuation of all treatment
  The goal of treatment of chronic hepatitis B
Safety | End of treatment 6 months off-treatment
  To evaluate the safety and tolerability of VIR-2218 in combination with peginterferon alfa-2a in non-cirrhotic adults with chronic HBV infection

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001606-DK.html